CLINICAL TRIAL: NCT03706755
Title: Comparison of Two Doses of Norepinephrine in Preventing Hypotension After Spinal Anesthesia for Cesarean Section
Brief Title: Comparison of Two Doses of Norepinephrine in Preventing Hypotension After Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben marzouk Sofiene, clinical associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Norepinephrine
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Adverse Effect; Hypotension; Cesarean Section Complications; Vasopressor
Keywords: spinal anesthesia; blood pressure; norepinephrine; Cesarean Section
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): group A: will receive 1 mcg/Kg of Norepinephrine intravenously
  Interventions: Drug: Norepinephrine: 1mcg/kg
- B (Active Comparator): group B: will receive 0.5 mcg/Kg of Norepinephrine intravenously
  Interventions: Drug: Norepinephrine 0,5mcg/kg

INTERVENTIONS:
Drug: Norepinephrine: 1mcg/kg — intervention:Parturients will receive Norepinephrine: a bolus of 1 mcg/Kg immediately after SA (preventive bolus) then they will receive complementary doses of Norepinephrine (half dose: 0.5 mcg/Kg) to maintain systolic blood pressure above 80 % of baseline
  Other Names: Noraline; Noradrenaline
  Arms: A
Drug: Norepinephrine 0,5mcg/kg — intervention: Parturients will receive Norepinephrine: a bolus of 0.5 mcg/Kg immediately after SA (preventive bolus) then they will receive complementary doses of Norepinephrine (half dose: 0.25 mcg/Kg) to maintain systolic blood pressure above 80 % of baseline
  Other Names: Noraline; Noradrenaline
  Arms: B

SUMMARY:
The purpose of the study is to determine the more effective intravenous bolus of norepinephrine for maintaining blood pressure during a spinal anesthesia for a cesarean delivery with the fewer side effects. Low blood pressure has been shown to decrease uterine perfusion and foetal outcomes during cesarean delivery under spinal anesthesia. For elective or semi-urgent cesarean delivery, all participants will receive spinal anesthesia with a local anesthetic and either sufentanil or fentanyl. This study plans to enroll 124 pregnant women. Patients will be randomly assigned according to a computer generated system to be in one of two groups.

DETAILED DESCRIPTION:
This study will be a prospective, randomized, active treatment controlled trial.

After written and informed consent, the study participants will be randomly assigned using a computer generated table to 1 of 2 treatment groups prior to cesarean delivery.

Group A will receive an intravenous bolus of 1mcg/Kg of norepinephrine bitartrate to maintain systolic blood pressure (SBP) within 80-120% of baseline before the spinal anesthesia.

Group B will receive an intravenous bolus of 0.5mcg/kg of norepinephrine bitartrate to maintain systolic blood pressure (SBP) within 80-120% of baseline before the spinal anesthesia.

Patients will be admitted to holding area. Baseline arterial blood pressure and heart rate will be measured in supine position, with left uterine displacement. Baseline blood pressure will be calculated as the mean of three consecutive SBP measurements taken 3 minutes apart. 500 mL of Lactated Ringer solution will be administered immediately after induction of spinal anesthesia at the outflow rate of 100ml per hour.

The primary endpoints are: the percentage of decrease of systolic blood pressure and mean blood pressure respectively measured by delta SBP and delta MBP before delivery ( difference between baseline and the lowest systolic and mean blood pressure respectively) and during cesarean delivery

The secondary endpoints are:

the timing of the first maternal hypotension (defined as a decrease of SBP >20% of baseline and/or PAS<100mmHg), duration of hypotension, incidence of hypotension, number of rescue boluses, norepinephrine consumption (mean dose of Norepinephrine to maintain blood pressure between 80 and 100 % of baseline values after the primary preventive bolus), maternal adverse effects and fetal outcomes.

Study participants will receive a standard spinal anesthetic consisting of 0.5% hyperbaric bupivacaine (2 mL) with either sufentanil (5 mcg) or fentanyl (50 mcg) at L3-4 or L4-5. Prior to surgical incision, the spinal sensory level will be tested to the bilateral T6-T4 dermatomal level. The patients will be positioned supine with a wedge placed under the right hip to avoid aortocaval compression. Both the patient and the researcher's assistant (who will collect data) will be blinded as to the administered Norepinephrine bolus A or B.

When PAS<80% of baseline or < 100 mmHg a bolus of Norepinephrine will be administrated(half dose A or B).

The study will end when cesarean section is completed and the patient transferred to the post-operative care unit.

Measured variables will include systolic, diastolic and mean non-invasive blood pressure, heart rate, number of rescue boluses and Norepinephrine consumption nausea and vomiting will be recorded whenever present during the surgical procedure as well as reactive hypertension (defined as a rise of SBP >20% of baseline or SBP>140mmHg) and arrhythmia. Bradycardia (HR less than 50 BPM) will be treated with Atropine 1mg IV.

Apgar score and fetal cord blood analysis (pH) at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Elective or semi-urgent CD under spinal anesthesia
* Age over 18 years
* Healthy singleton pregnancy beyond 36 weeks' gestation
* American Society of Anesthesiologists (ASA) physical status classification 2
* Weight 50 to 100 kg, and height 150 to 180 cm

Exclusion Criteria:

* Emergency CD red code ( extraction time <15 min)
* Allergy or hypersensitivity to norepinephrine or sulfite
* Preexisting or pregnancy-induced hypertension, preeclampsia, eclampsia, the use of cardiac medication or medication for blood pressure control
* multiple gestation
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities
* Suspicion of abnormal placentation
* History of diabetes mellitus (excluding gestational diabetes)
* Use of monoamine oxidase inhibitors, triptyline or imipramine antidepressants
* documented history of postoperative nausea and vomiting, previous gastric bypass surgery, history of chronic opioid use (chronic pain syndrome)
* Patient refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure variation before delivery | time from immediately after spinal anesthesia until delivery
  difference between the baseline systolic blood pressure (SBP0) and the lowest systolic blood pressure (SBPmin) registred before delivery and computed as (SBP min -SBP0)/SBP0
mean blood pressure variation before delivery | time from immediately after spinal anesthesia until delivery
  difference between the baseline mean blood pressure(MBP0) and the lowest mean blood pressure (MBPmin) registred before delivery and computed as (MBP min -MBP0)/MBP0
systolic blood pressure variation during cesarean delivery | time from immediately after spinal anesthesia until the end of surgery
  difference between the baseline systolic blood pressure (SBP0) and the lowest systolic blood pressure (SBPmin) registred during the cesarean section
mean blood pressure variation during cesarean delivery | time from immediately after spinal anesthesia until the end of surgery
  difference between the baseline mean blood pressure (MBP0) and the lowest systolic blood pressure (MBPmin) registred during the cesarean section

SECONDARY OUTCOMES:
Time to administartion of the first rescue bolus | time from immediately after spinal anesthesia until delivery
  timing of the first hypotension(defined as a decrease of SBP >20% of baseline and/or PAS<100mmHg) recsue bolus will be given at that moment
duration of hypotension | immediately after spinal anesthesia until the end of surgery
  duration of each episode of hypotension in minutes
number of rescue boluses | immediately after spinal anesthesia until the end of surgery
  the number of boluses to treat hypotension
Incidence of hypotension | tile from right after spinal anesthesia until delivery
  incidence of hypotension after the primary preventive bolus
Norepinephrine consumption | time fro right after spinal anesthesia until the end of surgery
  Mean dose of Norepinephrine ( micrograms) given to maintain blood pressure between 80 and 100 % of baseline values after the primary preventive bolus
Nausea | time of surgery (right after spinal anesthesia until end of surgery)
  Incidence of nausea. Measure will be done according to a simple scale: 0= no nausea; 1= nausea [Time
Vomiting | time of surgery (right after spinal anesthesia until end of surgery)
  incidence of Vomiting (V) during cesarean section with an infusion of a bolus Norepinephrine. Measure will be done according to a simple scale: 0= no vomiting; 1= vomiting
Bradycardia | immediately after spinal anesthesia until the end of surgery
  heart rate less than 50 BPM
arrhythmia | time of surgery (right after spinal anesthesia until end of surgery)
  incidence of arrhythmic events during cesarean section with an infusion of a bolus of Norepinephrine
Hypertension | right after spinal anesthesia until end of surgery)]
  a rise of systolic blood pressure (SBP)>20% of baseline or SBP>140mmHg
Apgar score | at time of birth
  apgar at 1 and 5 minutes Apgar at 1 and 5 minutes
mean pH of the fetal cord blood | time of birth
  Fetal cord blood analysis will be done immediately after delivery in order to determine the pH value ( ie : logarithm of the blood concentration of hydrogen ions H+)in each group

CONTACTS AND LOCATIONS:
Overall Officials: HAYEN Hayen maghrebi, professor, Study Chair — University Tunis El Manar
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia